CLINICAL TRIAL: NCT06662682
Title: Acute Effects of Whole-Body Vibration on Pain, Neuromuscular Performance and Gait Quality in Patients with Knee Osteoarthritis. a Randomized Controlled Trial.
Brief Title: Effects of Whole-Body Vibration in Patients with Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Wolfgang Kemmler, PhD, Head of Research, Friedrich-Alexander-Universität Erlangen-Nürnberg
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RadioSurg1
Record Dates: First submitted 2024-10-18; First posted 2024-10-29 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthristis
Keywords: Knee OA; whole-body vibration; pain; physical function; gait parameters
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor were unaware of participants status and were not allowed to ask correpondingly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whole-Body Vibration (Experimental): The intervention (IC) will be specified as a five-minute Whole-Body Vibration session.
  Interventions: Other: Whole-Body Vibration
- Control Condition (Other): The control condition (CC) will conduct the same protocol as the intervention condition. The only difference will be that the vibration plate will be switched off.
  Interventions: Other: Control Condition

INTERVENTIONS:
Other: Whole-Body Vibration — The intervention (IC) will be specified as a five-minute Whole-Body Vibration session. The WBV take place on a side alternating vibration plate (Wellengang, Germany). The patients stand barefoot on the vibration plate on a prescribed position. In this position the amplitude will be 6-7mm. The WBV protocol contains mobilizing sequences with lower frequencies and activating sequences with higher frequencies
  Arms: Whole-Body Vibration
Other: Control Condition — Non-intervention control condition
  Arms: Control Condition

SUMMARY:
Knee osteoarthritis is a chronic joint disease with an impact on quality of life and an increasing incidence what leads to huge costs and burden on the economy.

The present study investigates immediate effects of whole-body vibration on pain, neuromuscular performance, and gait quality in patients with knee osteoarthritis. Eligible patients (n=20) with knee osteoarthritis grade 2 or 3 on Kallgren Lawrence will complete a 5 minute WBV training and a control condition in a randomized order (cross over design). Pain, maximum strength of the leg flexors and extensors, the chair rise test and gait parameters will be measured directly before and after the intervention/control.

ELIGIBILITY:
Inclusion Criteria:

* x-ray confirmed knee osteoarthritis (Kallgren-Lawrence 2-3)
* knee pain (NRS 0-10 >2) for 3 months and at least 50% of the last 30 days

Exclusion Criteria:

* contraindications for WBV (acute injuries of the musculoskeletal system, new joint endoprosthesis, pregnancy, acute thrombosis, Epilepsia, cholecystolithiasis, nephrolithiasis, heart pace maker),
* other pathologies affecting gait or neuromuscular performance (rheumatic
* opioid medications, cortisol medications and intraarticular injections in the knee during the ist 3 months.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Changes in pain of the osteo-arthrotic knee | Changes in pain of the osteoarthrotic knee during the treadmill test as determined on a visual analogue scale (VAS 0-10) before and after 5 min of intervention
  Changes in pain of the osteo-arthrotic knee during the treadmill test as determined on a visual analogue scale (VAS 0-10).

SECONDARY OUTCOMES:
Changes in isometric maximum leg flexion strength of the osteoarthritis knee | Changes in isometric maximum leg flexion strength of the osteoarthritis knee before and after 5 min of Intervention.
  Changes in isometric maximum leg flexion strength of the osteoarthritis knee as determined by dynamometer (easy torque, Tonus, Germany)
Changes in isometric maximum leg extension strength of the osteoarthritis knee | Changes in isometric maximum leg extension strength of the osteoarthritis knee before and after 5 min of Intervention
  Changes in isometric maximum leg extension strength of the osteoarthritis knee as determined by dynamometer (easy torque, Tonus, Germany)
Changes of number of repetitions in the 30 s sit to stand (chair rise) test | Changes in number of repetitions in the 30 s sit-to-stand test before and after 5 min of intervention
  Changes in number of repetitions in the 30 s sit-to-stand test as suggested by Guralnik et al.
Changes of ipsilateral stride length | Changes of ipsilateral stride length (cm) at treadmill as determined by the 4D motion high-performance lab ( (Firma Diers Formetric, Germany) before and after 5 min of Intervention
  Changes of ipsilateral stride length (cm) at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany)
Changes of ipsilateral stride time | Changes of ipsilateral stride length (cm) at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany) before and after 5 min of intervention.
  Changes of ipsilateral stride length (cm) at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany)
Changes of stride width | Changes of stride width (cm) at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany) before and after 5 min of intervention.
  Changes of stride width (cm) at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany)
Changes of ipsilateral stance time | Changes of ipsilateral stance time (%) at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany) before and after 5 min of intervention
  Changes of ipsilateral stance time (%) at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany)
Changes of ipsilateral single support time | Changes of ipsilateral single support time (%) at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany) before and after 5 min of intervention
  Changes of ipsilateral single support time (%) at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany)
Changes of double support time | Changes of double support time (%) at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany) before and after 5 min of intervention
  Changes of double support time (%) at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany)
Changes of trunk inclination | Changes of trunk inclination (mm) at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany) before and after 5 min of intervention
  Changes of trunk inclination (mm) at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany)
Changes of ipsilateral und kontralateral knee angle in frontal plane | Changes of ipsilateral und kontralateral knee angle (°) in frontal plane at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany) before and after 5 min of intervention
  Changes of ipsilateral und kontralateral knee angle (°) in frontal plane at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany)
Changes of ipsilateral und kontralateral knee angle in sagital plane | Changes of ipsilateral und kontralateral knee angle in sagital plane (°) at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany) before and after 5 min of intervention
  Changes of ipsilateral und kontralateral knee angle in sagital plane (°) at treadmill as determined by the 4D motion high-performance lab (Firma Diers Formetric, Germany)

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Betsch, MD, Study Director — University Hospital Erlangen, Germany
Locations (1):
- Oniversity Hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] von Stengel S, Kemmler W, Engelke K, Kalender WA. Effect of whole-body vibration on neuromuscular performance and body composition for females 65 years and older: a randomized-controlled trial. Scand J Med Sci Sports. 2012 Feb;22(1):119-27. doi: 10.1111/j.1600-0838.2010.01126.x. Epub 2010 May 24. PMID 20500555